CLINICAL TRIAL: NCT00502086
Title: Efficacy and Safety of Viusid, a Nutritional Supplement, in Patients With Hepatic Cirrhosis Secondary to Hepatitis C Virus Infection. A Randomized, Controlled and Double Blind Study.
Brief Title: Efficacy and Safety of Viusid in Patients With Hepatic Cirrhosis Secondary to Hepatitis C Virus Infection.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Eduardo Vilar Gómez, National Institute of Gastroenterology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VIUHCV-07
Record Dates: First submitted 2007-07-13; First posted 2007-07-17 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Cirrhosis; Chronic Hepatitis C
Keywords: Chronic hepatitis C; Cirrhosis of the liver; Mortality; Complications; Health-related quality of live; Hepatocellular carcinoma; Nutritional supplement
MeSH Terms: conditions — Fibrosis; Hepatitis C, Chronic; Carcinoma, Hepatocellular | interventions — Viusid; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental): Viusid, three sachets daily during 96 weeks
  Interventions: Dietary Supplement: Viusid (nutritional supplement)
- 2 (Placebo Comparator): Placebo three sachets daily during 96 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Viusid (nutritional supplement) — Viusid three sachets daily during 96 weeks
  Other Names: Nutritional supplement
  Arms: I
Other: Placebo — Placebo three sachets daily during 96 weeks
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate whether Viusid, a nutritional supplement, reduce the mortality and the complications (ascites, spontaneous bacterial peritonitis, hepatorenal syndrome, hepatic encephalopathy, gastrointestinal bleeding, sepsis and hepatocellular carcinoma) of patients with cirrhosis of the liver secondary to HCV infection in comparison with placebo, during 96 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histological or clinical diagnosis of cirrhosis.
* HCV infection confirmed on a positive test for anti-HCV antibody and HCV RNA detectable in serum by Polymerase Chain Reaction.
* Patients who were non-responders to previous treatment with pegylated interferon and ribavirin or naïve patients with decompensated cirrhosis (Child-Pugh score ≥ 7) who had contraindicated the antiviral treatment.
* Presence of compensated or decompensated (Stage A, B or C according to the Child-Pugh Classification).
* Absence of clinical and ultrasonographic evidence of liver cancer, with α-fetoprotein levels ≤ 200 ng/ml.

Exclusion Criteria:

* Age less than 18 or greater than 70 years.
* Presence of uncontrollable clinical or biochemical complications related to severe liver failure (hepatic encephalopathy, hepatorenal syndrome, gastrointestinal bleeding, serum bilirubin level greater than 5 mg/dL, international normalized ratio greater than 2.5).
* Active alcoholism.
* Serum creatinine greater than 2 mg/dL.
* Hepatocellular carcinoma.
* Refusal to participate in the study.
* Concomitant disease with reduced life expectancy.
* Severe psychiatric conditions.
* Co-infection with hepatitis A or B or HIV.
* Drug dependence.
* Pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The mortality secondary to liver failure at 96 weeks. | 96 weeks

SECONDARY OUTCOMES:
The complication rates during the treatment. The hepatitis-related quality of live during the treatment. Clinical Activity Index during the treatment. The hepatocellular carcinoma incidence during the treatment. | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Vilar Gómez, PhD, Principal Investigator — National Institute of Gastroenterology, Havana, Cuba
Locations (1):
- National Institute of Gastroenterology, Plaza de la Revolución, La Habana, Cuba

REFERENCES:
- [Background] Vilar Gomez E, Gra Oramas B, Soler E, Llanio Navarro R, Ruenes Domech C. Viusid, a nutritional supplement, in combination with interferon alpha-2b and ribavirin in patients with chronic hepatitis C. Liver Int. 2007 Mar;27(2):247-59. doi: 10.1111/j.1478-3231.2006.01411.x. PMID 17311621
- [Derived] Vilar Gomez E, Sanchez Rodriguez Y, Torres Gonzalez A, Calzadilla Bertot L, Arus Soler E, Martinez Perez Y, Yasells Garcia A, Abreu Vazquez Mdel R. Viusid, a nutritional supplement, increases survival and reduces disease progression in HCV-related decompensated cirrhosis: a randomised and controlled trial. BMJ Open. 2011 Jan 1;1(2):e000140. doi: 10.1136/bmjopen-2011-000140. PMID 22021873